CLINICAL TRIAL: NCT00167557
Title: Tacrolimus Monotherapy in OLT Recipients With HCV Under Preemptive Treatment With Interferon and Ribavirin
Brief Title: Orthotopic Liver Transplant (OLT) Recipients With Hepatitis C Virus (HCV) Under Preemptive Treatment
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The PI left the institution.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-04-0346; Astellas Pharma; FHIprojectno.JK-04-002
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Hepatitis C
Keywords: Liver Transplantation
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm Study (Experimental)
  Interventions: Drug: Pegylated Interferon; Drug: Ribavirin; Procedure: Liver Biopsy

INTERVENTIONS:
Drug: Pegylated Interferon — 180mcg SC weekly starting 30 days post transplant
Drug: Ribavirin — goal dose 13mg/kg starting 120 days post transplant for a minimum of 48 wks
Procedure: Liver Biopsy — Liver biopsies performed at 9 points in time from time of liver transplant

SUMMARY:
After a liver transplant, the hepatitis C virus (which destroyed one's own liver) eventually comes back. In many patients, this will eventually cause the loss of the new liver and can also confuse the doctors taking care of them because it is hard to tell the difference between one's body rejecting the new liver and hepatitis. This can cause serious treatment errors that can lead to more severe hepatitis or to rejection of the liver. Some of the drugs used to prevent rejection of one's new liver can cause the hepatitis to come back in a more severe form. This is especially true for the drugs known as corticosteroids.

Right now, the only effective treatment against hepatitis C is a combination of two drugs called interferon and ribavirin. These drugs act by strengthening one's immune system to fight the virus and by directly reducing the reproduction of the virus. Because the treatment with these drugs is associated with many side effects, there is little experience with treating patients after liver transplantation with them.

In the investigators' transplant program, they have decided to treat all patients with hepatitis C as early as possible after transplantation and to follow them closely for the development of hepatitis and side effects of the treatment. The investigators treat one's hepatitis as early as possible, before any actual damage has occurred in the new liver. This approach has been tried before but it has been hard to tell if it has worked or not. The main reason for failure was that many patients could not complete the treatment due to side effects. The investigators' purpose is to treat those side effects aggressively so that most patients can complete the treatment course.

The purpose of this study is to collect all the data regarding the investigators' treatment protocol so that they will be able to learn if this form of treatment is beneficial.

The study includes performing liver biopsies at scheduled times after one's liver transplant and for scheduled blood tests to see how much virus is still in the blood. If patients show signs that they are not responding to treatment they will be removed from the study.

DETAILED DESCRIPTION:
HCV recurs in the transplanted liver almost invariably. The clinical course is variable and ranges from no hepatitis to severe aggressive hepatitis with cirrhosis. Factors that affect outcome are high viral load prior to OLT, genotype, and immunosuppressive regimen. Recent studies indicate that the severity of recurrence is increasing with longer follow up, and longevity of both graft and patient is compromised by HCV. Viral load appears to be particularly affected by corticosteroids. The impact of mycophenolate mofetil and tacrolimus is not certain. The results of re-transplantation are generally poor and seem to be a non-cost beneficial way to deal with recurrence HCV cirrhosis. Additionally, re-transplantation deprives other patients from getting OLT in a timely fashion.

Recent studies have shown that with intensive alpha interferon and ribavirin treatment, up to 40% of patients can be cleared of virus as measured by PCR. Thus, despite the cost and side effects of this treatment, it appears justified to treat recurrence preemptively.

Due to the deleterious effects of high dose Corticosteroids it seems logical to attempt to withdraw them as soon as possible from treatment. MMF is often incompatible with interferon and ribavirin treatment due to leukopenia and anemia. The same is true for sirolimus. Thus, most patients will eventually be treated with Tacrolimus monotherapy. Presently, numerous patients end up being treated with Tacrolimus monotherapy as part of the reduction in immune suppression, which occurs over time. There is, however, very little prospective data regarding Tacrolimus monotherapy and almost no data on the specific issue of monotherapy in HCV patients. Even less is known with respect to this type of treatment while using interferon and ribavirin.

Our purpose in this protocol is to examine both the effect of preemptive antiviral treatment on recurrent HCV and the effect of Tacrolimus monotherapy in this setting. This may be important as more and more programs are turning to preemptive anti viral treatment and the issue of appropriate immune suppression becomes seminal to this discussion.

Aims

1. To determine the safety and efficacy of PEG interferon and ribavirin in the treatment of HCV recurrence after OLT.
2. To determine the effectiveness and safety of maintenance dose of PEG interferon to delay progression of fibrosis and histologic damage, in non-responders to the initial regimen of PEG interferon and ribavirin.
3. To determine the effect of early prednisone withdrawal in the rate of response to treatment with PEG interferon and ribavirin.
4. To assess the feasibility of Tacrolimus monotherapy in patients undergoing treatment for HCV recurrence post transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patients between 18 and 70 years of age
2. All liver transplant patients with a positive HCV RNA by PCR within 30 days after transplant.
3. No evidence of acute or chronic rejection within 4 weeks of enrollment
4. Compensated liver disease according to the following criteria:

   * Hemoglobin > 10 gm/dL;
   * Neutrophil count > 1,000/mm3;
   * Platelet count > 50,000/mm3;
   * Serum creatinine < 2.0 mg/dL.
5. Documentation of adequate contraception in females and males sexually active or of childbearing potential.

Exclusion Criteria:

1. Hypersensitivity to alpha interferon and/or ribavirin
2. Previous treatment with interferon and/or ribavirin post liver transplantation
3. HIV
4. Autoimmune hepatitis
5. Active alcohol or substance abuse
6. Non compliance
7. Hemoglobinopathies or hemolytic anemia
8. Clinical significant retinal abnormalities
9. Decompensated cardio-vascular, endocrine, pulmonary, renal, immune, metabolic, dermatologic or psychiatric illness
10. Re-transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Viral clearance after liver transplantation | 3 yrs. post liver transplant

SECONDARY OUTCOMES:
histological progression of fibrosis and inflammation | 3 yrs. post liver transplant
rate of rejection on HCV treatment | 3 yrs post liver transplant

CONTACTS AND LOCATIONS:
Overall Officials: Hadar J Merhav, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States